CLINICAL TRIAL: NCT02471716
Title: A Phase 1/2 Study of Cabiralizumab, an Anti-CSF1 Receptor Antibody, in Patients With Pigmented Villonodular Synovitis (PVNS)/ Diffuse Type Tenosynovial Giant Cell Tumor (Dt-TGCT)
Brief Title: Study of Cabiralizumab in Patients With Pigmented Villonodular Synovitis / Diffuse Type Tenosynovial Giant Cell Tumor
Acronym: FPA008-002
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Five Prime Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPA008-002
Record Dates: First submitted 2015-06-01; First posted 2015-06-15 (Estimated); Results first posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2020-07

CONDITIONS: Pigmented Villonodular Synovitis; Tenosynovial Giant Cell Tumor
Keywords: Diffuse Type Tenosynovial Giant Cell Tumor (dt-TGCT)
MeSH Terms: conditions — Synovitis, Pigmented Villonodular; Giant Cell Tumor of Tendon Sheath | interventions — cabiralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1 FPA008 Dose Escalation (Experimental): IV infusion; safety data will be reviewed prior to dose escalation decision. Dose escalation will complete when recommended dose (RD) is determined. RD will be the maximum tolerated dose or lower dose that provide adequate PK exposure and biologic activity with tolerability.
  Interventions: Biological: FPA008
- Phase 2 FPA008 Dose Expansion (Experimental): IV infusion; once MTD and/or RD has been determined in Phase 1, expansion cohorts of approximately 30 patients (each cohort) with PVNS or dt-TGCT will be enrolled to characterize clinical activity and safety profile of the RD. Treatment is planned to continue for up to 24 weeks or 56 weeks.
  Interventions: Biological: FPA008

INTERVENTIONS:
Biological: FPA008 — FPA008 will be administered by IV infusion over approximately 30 minutes every 2 or 4 weeks
  Other Names: Cabiralizumab

SUMMARY:
This is a phase 1/2 single arm, open-label, safety, tolerability, and PK study of cabiralizumab in PVNS/dt-TGCT patients.

DETAILED DESCRIPTION:
A Phase 1/2 study was an open-label, dose escalation and dose expansion study designed to evaluate the pharmacokinetics, pharmacodynamics, safety and preliminary efficacy of cabiralizumab, a CSF1-R monoclonal antibody, inpatients with unresectable diffuse tenosynovial giant cell tumors (TGCT).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of inoperable PVNS/ dt-TGCT or potentially resectable tumor that would result in unacceptable functional loss or morbidity as determined by a qualified surgeon or multi-disciplinary tumor board (must be documented in the CRF during screening)
* Measurable PVNS/dt-TGCT by RECIST 1.1 on MRI
* ECOG performance status <1

Exclusion Criteria:

* Prior therapy with an anti-CSF1R antibody
* Prior therapy with PLX3397 unless discontinued for intolerance (i.e., non-progression on prior kinase inhibitor)
* Liver function tests (including ALT, AST, and total bilirubin), outside of the range of local laboratory normal at Screening
* Inadequate organ or bone marrow function
* History of congestive heart failure or myocardial infarction <1 year prior to first study dose administration
* Significant abnormalities on ECG at Screening
* Contraindications to MRI and use of intravenous gadolinium-based contrast agents
* Creatine Kinase ≥ 1.5x the upper limit of normal
* Positive test for latent TB at Screening (Quantiferon test)
* Active known or suspected autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Lead, Study Director — Five Prime Therapeutics, Inc.
Locations (12):
- United States (5):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sarcoma Oncology Research Center LLC, Santa Monica, California
  - Stanford Medicine, Stanford, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
- France (2):
  - Institut Bergonie- CRLCC de Bordeaux et du Sud-Ouest, Bordeaux
  - Centre Léon Bérard, Lyon
- Leiden University Medical Center, Leiden, Netherlands
- Klinika Nowotworow Tkanek Miekkich, Kosci i Czerniakow, Centrum Onkologii-Instytut im. M. Sklodowskiej-Curie, Warsaw, Poland
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Oxford University Hospital NHS Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 FPA008 Dose Escalation 1mg/kg: Dose Escalation cohort: Dose level 1: 1 mg/kg cabiralizumab every 2 weeks
- Phase 1 FPA008 Dose Escalation 2mg/kg: Dose Escalation cohort: Dose level 2: 2 mg/kg cabiralizumab every 2 weeks
- Phase 1 FPA008 Dose Escalation 4mg/kg: Dose Escalation cohort: Dose level 3: 3 mg/kg cabiralizumab every 2 weeks
- Phase 2 FPA008 Dose Expansion Cohort 2A: Dose Expansion Cohort: patients were treated with 4 mg/kg cabiralizumab every 2 weeks in 28-day cycles for up to 12 doses.
- Phase 2 FPA008 Dose Expansion Cohort 2B: Dose Expansion Cohort: patients were treated with 4 mg/kg cabiralizumab on Cycle 1 Day 1 and Cycle 1 Day 15 then every 4 weeks thereafter for up to 12 months after Cycle 1, Day 1.
Period: Overall Study
Arm/Group | Phase 1 FPA008 Dose Escalation 1mg/kg | Phase 1 FPA008 Dose Escalation 2mg/kg | Phase 1 FPA008 Dose Escalation 4mg/kg | Phase 2 FPA008 Dose Expansion Cohort 2A | Phase 2 FPA008 Dose Expansion Cohort 2B
Started | 3 | 3 | 3 | 33 | 24
Completed | 3 | 2 | 3 | 18 | 8
Not Completed | 0 | 1 | 0 | 15 | 16
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2 | 5
Not completed — Study Terminiated by sponsor | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 FPA008 Dose Escalation 1mg/kg | Phase 1 FPA008 Dose Escalation 2mg/kg | Phase 1 FPA008 Dose Escalation 4mg/kg | Phase 2 FPA008 Dose Expansion Cohort 2A | Phase 2 FPA008 Dose Expansion Cohort 2B | Total
Number analyzed (Participants) | 3 | 3 | 3 | 33 | 24 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 3 | 32 | 22 | 62
  >=65 years | 0 | 1 | 0 | 1 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (11.24) | 40.7 (23.07) | 41.7 (7.51) | 38 (12.77) | 44.1 (15.32) | 40.8 (14.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 23 | 10 | 40
  Male | 0 | 0 | 2 | 10 | 14 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Black | 0 | 0 | 0 | 0 | 2 | 2
  Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 2 | 9 | 9 | 25
  Asian | 0 | 1 | 0 | 5 | 1 | 7
  Other | 0 | 0 | 0 | 19 | 8 | 27
  Unknown | 0 | 0 | 1 | 0 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Grade 3 and Grade 4 Adverse Events (AEs) and Defined as Dose-limiting Toxicities (DLTs) in Phase 1
Description: Number of participants with grade 3 and grade 4 adverse events (AE) defined as dose limiting toxicities (DLTs) in Phase 1
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 FPA008 Dose Escalation 1mg/kg | Phase 1 FPA008 Dose Escalation 2mg/kg | Phase 1 FPA008 Dose Escalation 4mg/kg
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

2. Primary Outcome: The Incidence of Investigator-assessed, Confirmed Objective Responses (ORR) Per RECIST 1.1 (Phase 2)
Description: Number of confirmed objective responses (ORR) as assessed by the investigator per RECIST 1.1 (Phase 2)
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 FPA008 Dose Expansion Cohort 2A | Phase 2 FPA008 Dose Expansion Cohort 2B
Number analyzed (Participants) | 32 | 24
Participants | 8 | 8

3. Secondary Outcome: PK Parameters of Cabiralizumab: Area Under Concentration-time Curve (AUC)
Description: Area under serum concentration-time curve (AUC) for cabiralizumab as a PK parameter
Time Frame: 52 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug x day/mL
Arm/Group | Phase 1 FPA008 Dose Escalation 1mg/kg | Phase 1 FPA008 Dose Escalation 2mg/kg | Phase 1 FPA008 Dose Escalation 4mg/kg | Phase 2 FPA008 Dose Expansion Cohort 2A | Phase 2 FPA008 Dose Expansion Cohort 2B
Number analyzed (Participants) | 3 | 2 | 1 | 2 | 3
ug x day/mL | 102 (10.2) | 283 (26.3) | 593 (31.3) | 660 (17.7) | 593 (12.6)

4. Secondary Outcome: Maximum Serum Concentration (Cmax).
Description: Composite PK parameters of cabiralizumab: Maximum observed serum concentration
Time Frame: 52 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Phase 1 FPA008 Dose Escalation 1mg/kg | Phase 1 FPA008 Dose Escalation 2mg/kg | Phase 1 FPA008 Dose Escalation 4mg/kg | Phase 2 FPA008 Dose Expansion Cohort 2A | Phase 2 FPA008 Dose Expansion Cohort 2B
Number analyzed (Participants) | 3 | 3 | 3 | 30 | 24
ug/mL | 22.5 (14.3) | 52.1 (22) | 91.2 (15) | 91.8 (24.8) | 87 (12.6)

5. Secondary Outcome: Minimum Serum Concentration (Cmin).
Description: Composite PK parameters of cabiralizumab: minimum serum concentration (Cmin).
Time Frame: 52 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Phase 1 FPA008 Dose Escalation 1mg/kg | Phase 1 FPA008 Dose Escalation 2mg/kg | Phase 1 FPA008 Dose Escalation 4mg/kg | Phase 2 FPA008 Dose Expansion Cohort 2A | Phase 2 FPA008 Dose Expansion Cohort 2B
Number analyzed (Participants) | 3 | 3 | 3 | 30 | 24
ug/mL | 2.18 (117) | 7.26 (41.8) | 21.2 (59.2) | 23.9 (38.3) | 22.6 (28.2)

6. Secondary Outcome: Pharmacokinetic Clearance (CL).
Description: Composite PK parameters of cabiralizumab: clearance (CL)
Time Frame: 52 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/d
Arm/Group | Phase 1 FPA008 Dose Escalation 1mg/kg | Phase 1 FPA008 Dose Escalation 2mg/kg | Phase 1 FPA008 Dose Escalation 4mg/kg | Phase 2 FPA008 Dose Expansion Cohort 2A | Phase 2 FPA008 Dose Expansion Cohort 2B
Number analyzed (Participants) | 3 | 2 | 1 | 2 | 3
L/d | .663 (16.6) | .416 (24.5) | .694 (0) | .307 (44.9) | .525 (8.42)

7. Secondary Outcome: The Incidence of AEs.
Description: treatment-emergent adverse events (TEAEs) by incidence for the Safety Population. Patients with at lease 1 TEAE.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 FPA008 Dose Escalation 1mg/kg | Phase 1 FPA008 Dose Escalation 2mg/kg | Phase 1 FPA008 Dose Escalation 4mg/kg | Phase 2 FPA008 Dose Expansion Cohort 2A | Phase 2 FPA008 Dose Expansion Cohort 2B
Number analyzed (Participants) | 3 | 3 | 3 | 33 | 24
Participants | 3 | 3 | 3 | 33 | 24

8. Secondary Outcome: The Incidence of Clinical Laboratory Abnormalities.
Description: The number of patients with a clinical laboratory that is outside the normal range at some time point during the study
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | Phase 1 FPA008 Dose Escalation 1mg/kg | Phase 1 FPA008 Dose Escalation 2mg/kg | Phase 1 FPA008 Dose Escalation 4mg/kg | Phase 2 FPA008 Dose Expansion Cohort 2A | Phase 2 FPA008 Dose Expansion Cohort 2B
Number analyzed (Participants) | 3 | 2 | 3 | 33 | 24
participants | 3 | 2 | 3 | 33 | 24

9. Secondary Outcome: The Incidence of ECG Abnormalities.
Description: The number of patients who had a change in their ECG that were clinically significant
Time Frame: 52 weeks
Population: The changes in the ECG parameters were not clinically significant in any dosing cohort in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 FPA008 Dose Escalation 1mg/kg | Phase 1 FPA008 Dose Escalation 2mg/kg | Phase 1 FPA008 Dose Escalation 4mg/kg | Phase 2 FPA008 Dose Expansion Cohort 2A | Phase 2 FPA008 Dose Expansion Cohort 2B
Number analyzed (Participants) | 3 | 3 | 3 | 33 | 24
Participants | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Duration of Response Per RECIST 1.1 in Phase 2
Description: The length of response per RECIST 1.1 from the time of first response to progression or going off study in Phase 2
Time Frame: 52 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 FPA008 Dose Expansion Cohort 2A | Phase 2 FPA008 Dose Expansion Cohort 2B
Number analyzed (Participants) | 8 | 8
months | 4.4 [3.2 to NA] — the upper bound of the confidence interval was not reached | NA [11.5 to NA] — The median duration of response was not reached

ADVERSE EVENTS:
Time Frame: Event reporting commences at the time of signing the informed consent. A treatment-emergent AE was defined as an AE that began or worsened in severity after at least 1 dose of study drug had been administered. Adverse event reporting continued through the End-of-Treatment Follow-Up Period or until 90 days (± 7 days) after the last dose of study drug, the patient underwent local therapy (e.g., resection, radiation) or a new systemic therapy was initiated.
Arm/Group | Phase 1 FPA008 Dose Escalation 1mg/kg | Phase 1 FPA008 Dose Escalation 2mg/kg | Phase 1 FPA008 Dose Escalation 4mg/kg | Phase 2 FPA008 Dose Expansion Cohort 2A | Phase 2 FPA008 Dose Expansion Cohort 2B
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 1/32 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 2/3 | 8/33 | 6/24
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 33/33 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 FPA008 Dose Escalation 1mg/kg (N=3) | Phase 1 FPA008 Dose Escalation 2mg/kg (N=3) | Phase 1 FPA008 Dose Escalation 4mg/kg (N=3) | Phase 2 FPA008 Dose Expansion Cohort 2A (N=33) | Phase 2 FPA008 Dose Expansion Cohort 2B (N=24)
Abdominal pain (Gastrointestinal disorders) | NA | NA | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | NA | NA | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | NA | NA | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | NA | NA | 0 | 0 | 1
Pyrexia (General disorders) | NA | NA | 0 | 1 | 1
Influenza like illness (General disorders) | NA | NA | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | NA | NA | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | NA | NA | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | NA | NA | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | NA | NA | 0 | 0 | 1
Viral infection (Infections and infestations) | NA | NA | 0 | 1 | 0
Cerebellar infarction (Nervous system disorders) | NA | NA | 0 | 1 | 0
Migraine (Nervous system disorders) | NA | NA | 0 | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | NA | NA | 0 | 0 | 1
Skin atrophy (Skin and subcutaneous tissue disorders) | NA | NA | 0 | 1 | 0
Twin reversed arterial perfusion sequence malformation (Congenital, familial and genetic disorders) | NA | NA | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | NA | NA | 0 | 1 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | NA | NA | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | NA | NA | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | NA | NA | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | NA | NA | 1 | 0 | 0
Endocarditis (Infections and infestations) | NA | NA | 1 | 0 | 0
Myocarditis (Cardiac disorders) | NA | NA | 0 | 2 | 0
Hypertension (Vascular disorders) | NA | NA | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 FPA008 Dose Escalation 1mg/kg (N=3) | Phase 1 FPA008 Dose Escalation 2mg/kg (N=3) | Phase 1 FPA008 Dose Escalation 4mg/kg (N=3) | Phase 2 FPA008 Dose Expansion Cohort 2A (N=33) | Phase 2 FPA008 Dose Expansion Cohort 2B (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Abnormal sensation in eye (Eye disorders) | 1 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 1
Conjunctival oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 2 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 6 | 7
Eyelid rash (Eye disorders) | 0 | 1 | 0 | 0 | 1
Eyelid skin dryness (Eye disorders) | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 4 | 5
Periorbital oedema (Eye disorders) | 2 | 2 | 2 | 20 | 13
Photophobia (Eye disorders) | 0 | 0 | 0 | 2 | 0
Scleritis (Eye disorders) | 0 | 0 | 0 | 2 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 3 | 5
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 5 | 3
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 4 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lip oedema (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 7 | 5
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 1
Face oedema (General disorders) | 0 | 1 | 2 | 22 | 12
Fatigue (General disorders) | 2 | 1 | 3 | 11 | 8
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 1 | 1
Local swelling (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1 | 1
Oedema (General disorders) | 0 | 0 | 0 | 1 | 2
Oedema peripheral (General disorders) | 2 | 1 | 2 | 19 | 8
Pain (General disorders) | 0 | 0 | 0 | 2 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 1 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 5 | 1
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 1 | 0
Swelling (General disorders) | 0 | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 6 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 10 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 4 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 3 | 21 | 16
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 4 | 3
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 7 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 10 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 7 | 3
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 3 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 5 | 2
Poor quality sleep (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 2
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2 | 4
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5 | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 17 | 13
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 5 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 11 | 10
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 8 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 5 | 1
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 3
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 4 | 5
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT02471716/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT02471716/SAP_001.pdf